CLINICAL TRIAL: NCT01233453
Title: Comparison of the Everolimus Eluting (XIENCE-V®, XIENCE-Prime® or PROMUS® Stent) With the Biolimus A9 Eluting NOBORI® Stent in All-comers: a Randomized Open Label Study
Brief Title: Comparison of the Everolimus Eluting With the Biolimus A9 Eluting Stent
Acronym: COMPARE-II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL25754.101.08
Record Dates: First submitted 2010-10-28; First posted 2010-11-03 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the everolimus eluting ® stent (Active Comparator): the everolimus eluting XIENCE-V®, XIENCE-Prime® or PROMUS® stent
  Interventions: Device: the everolimus eluting ® stent
- Biolimus A9 stent (Active Comparator): the Biolimus A9 eluting NOBORI® stent
  Interventions: Device: the Biolimus A9 eluting NOBORI® stent

INTERVENTIONS:
Device: the everolimus eluting ® stent — stenting in coronary artery disease using the XIENCE-V®, XIENCE-Prime® or PROMUS® stent
  Arms: the everolimus eluting ® stent
Device: the Biolimus A9 eluting NOBORI® stent — stenting in coronary artery disease using the Biolimus A9 eluting NOBORI® stent
  Arms: Biolimus A9 stent

SUMMARY:
This is a prospective, randomized, multi center study. Approximately 2700 patients will be entered in the study and will be randomized on a 2:1 basis. Patients who meet the eligibility criteria will be randomized to the everolimus eluting XIENCE-V®, XIENCE-Prime® or PROMUS® stent versus the Biolimus A9 eluting NOBORI® stent. Patients will be followed for 5 years.

DETAILED DESCRIPTION:
The main objective of the study is a head to head comparison of the everolimus eluting XIENCE-V ®, XIENCE-Prime® or PROMUS ® stent with the biolimus A9 eluting NOBORI® stent in order to observe whether there is a difference in clinical outcome between both stents in a real world / all-comer situation.

Clinical outcome of both stents will be assessed by the composite end point of: cardiac death, non fatal myocardial infarction and target vessel revascularization.

Endpoints

The primary end point of the study is the composite of safety (cardiac death, non fatal myocardial infarction) and efficacy (target vessel revascularization) at 12 months.

The secondary end points of the study are:

A) The combined endpoint of cardiac death, non fatal myocardial infarction, ischemic driven target lesion revascularization (TLR) rate at 12 months follow-up.

B) Incidence of Cardiac Death and Post-Procedural (>48h) MI rate at 12 months, 3 and 5 years C) Target lesion revascularization at 12 months, 3 and 5 years D) The combined endpoint of cardiac death, non fatal myocardial infarction, target vessel revascularization (TVR) rate at 3 and 5 years follow-up.

E) The combined endpoint of cardiac death, non fatal myocardial infarction and target vessel revascularization at 12 months, 3 and 5 years in STEMI patients, small vessels (< 2.75 mm RVD), long lesions (> 20 mm), female patients, DM patients and octogenarians. F) Procedural performance at the index procedures, measured by the ability to cross the lesions with the designated DES stent.

G) Incidence of definite and probable stent thrombosis at 12 months, 3 and 5 years time.

H) Incidence of definite, probable and possible stent thrombosis at 12 months, 3 and5 years time.

Overview of the study

This is a prospective, randomized, multi center study. Approximately 2700 patients will be entered in the study and will be randomized on a 2:1 basis. Patients who meet the eligibility criteria will be randomized to the everolimus eluting XIENCE-V®, XIENCE-Prime® or PROMUS® stent versus the Biolimus A9 eluting NOBORI® stent. Patients will be followed for 5 years.

The study population will consist of approximately 2700 patients (1 year enrollment of consecutive all-comers referred for percutaneous coronary intervention (PCI) with coronary artery or by-pass grafts lesions). Patients must meet all eligibility criteria for inclusion into the study.

Randomization will be performed by using a closed envelope with code N for the NOBORI stent and code E for the Everolimus eluting stent. Duration of the study The enrollment phase will start January 2009 and will stop December 2010. The followup phase will last till December 2015.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years old and has a life expectancy of 5 years.
2. Patient undergoes a PCI procedure for indications according to the Dutch and European guidelines
3. Patient is willing to comply with the extended follow-up period of 2 to 5 years(for secondary endpoint only)
4. Reference lumen diameter of the treated vessels between 2.0 - 4.0 mm.
5. Informed consent

Exclusion Criteria:

1. Expected non-adherence to dual antiplatelet therapy for 1 year (e.g: known allergy to ASA or thienopyridines like clopidogrel)
2. Expected major surgery within 30 days (these patients will receive bare metal stents)
3. Cardiogenic shock (Kilip class 4)
4. Previous PCI procedures with implantation of drug eluting stents within 1 year.
5. Expected loss for follow up
6. Enrollment in an investigative stent study with different stents
7. Inability to implant Nobori or Xience-V / Promus stent(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse coronary events | 12 months
  composite of cardiac death, non fatal myocardial infarction and target vessel revascularization

SECONDARY OUTCOMES:
Major adverse coronary events | 12 months
  The combined endpoint of cardiac death, non fatal myocardial infarction, ischemic driven target lesion revascularization (TLR) rate at 12 months follow-up.
Safety of stenting with drug eluting stents | 5 years
  Incidence of Cardiac Death and Post-Procedural (>48h) MI rate at 12 months, 3 and 5 years
Target lesion revascularization | 5 years
  Target lesion revascularization at 12 months, 3 and 5 years
Late major adverse coronary events | 5 years
  The combined endpoint of cardiac death, non fatal myocardial infarction, target vessel revascularization (TVR) rate at 3 and 5 years follow-up.
Major adverse coronary events in subgroups | 5 years
  The combined endpoint of cardiac death, non fatal myocardial infarction and target vessel revascularization at 12 months, 3 and 5 years in STEMI patients, small vessels (< 2.75 mm RVD), long lesions (> 20 mm), female patients, DM patients and octogenarians
Procedural performance | 1 year
  Procedural performance at the index procedures, measured by the ability to cross the lesions with the designated DES stent.
Stent Thrombosis | 5 years
  Incidence of definite and probable stent thrombosis at 12 months, 3 and 5 years time.
  Incidence of definite, probable or possible stent thrombosis at 12 months, 3 and 5 years time

CONTACTS AND LOCATIONS:
Overall Officials: Pieter C Smits, MD, PHD, Principal Investigator — Maasstad Ziekenhuis; A Serra, MD, Study Chair — Hospital del Mar; A J van Boven, MD, PHD, Study Chair — Medisch Centrum Leeuwarden; J J Goy, MD, Study Chair — Hopital Cantonal de Fribourg; V Voudris, MD, Study Chair — Onassis Heart Centre, Athens
Locations (11):
- Onassis cardiac Surgery Centre, Athens, Greece
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amphia Ziekenhuis, Breda
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maasstad Hospital, Rotterdam
- Spain (4):
  - Complejo Hospitalario Universitario Juan Canalejo, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Virgen Arrixaca, Murcia
  - Hospital Clinico universitario de Santiago de Compostella, Santiago de Compostela
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - Hopital Cantonal de Fribourg, Fribourg

REFERENCES:
- [Derived] Vlachojannis GJ, Smits PC, Hofma SH, Togni M, Vazquez N, Valdes M, Voudris V, Puricel S, Slagboom T, Goy JJ, den Heijer P, van der Ent M. Long-term clinical outcomes of biodegradable polymer biolimus-eluting stents versus durable polymer everolimus-eluting stents in patients with coronary artery disease: three-year follow-up of the COMPARE II (Abluminal biodegradable polymer biolimus-eluting stent versus durable polymer everolimus-eluting stent) trial. EuroIntervention. 2015 Jul;11(3):272-9. doi: 10.4244/EIJV11I3A53. PMID 26196753
- [Derived] Smits PC, Hofma S, Togni M, Vazquez N, Valdes M, Voudris V, Slagboom T, Goy JJ, Vuillomenet A, Serra A, Nouche RT, den Heijer P, van der Ent M. Abluminal biodegradable polymer biolimus-eluting stent versus durable polymer everolimus-eluting stent (COMPARE II): a randomised, controlled, non-inferiority trial. Lancet. 2013 Feb 23;381(9867):651-60. doi: 10.1016/S0140-6736(12)61852-2. Epub 2013 Jan 30. PMID 23374650